CLINICAL TRIAL: NCT02168933
Title: Randomized Controlled Trial of 308 nm Excimer Laser for Treatment of Nail Psoriasis
Brief Title: 308nm Excimer Laser for Treatment of Fingernail Psoriasis
Acronym: NAPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: American Society for Dermatologic Surgery (Other)
Responsible Party: Principal Investigator, Kristina Callis, M.D., University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FP00004323; 10032937 (Other: University of Utah OSP)
Record Dates: First submitted 2014-06-18; First posted 2014-06-20 (Estimated); Results first posted 2019-08-20 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Nail Psoriasis
Keywords: psoriasis; nail; laser; excimer; treatment
MeSH Terms: conditions — Psoriasis | interventions — Lasers, Excimer

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active excimer laser (Experimental): 308 nm excimer laser treatment: treatment with the laser by a dose protocol with increasing output.
  Interventions: Device: 308 nm excimer laser
- Sham excimer laser (Sham Comparator): Sham 308 nm excimer laser treatment: laser dose was administered with a cap that blocks all active UV passing through the device, therefore is a placebo, but because the procedure is the same, maintains a blind.
  Interventions: Device: Sham laser

INTERVENTIONS:
Device: 308 nm excimer laser — Biweekly treatments with 308 nm excimer laser for a total of 8 weeks
  Arms: active excimer laser
Device: Sham laser — Sham laser treatment to the control side biweekly for a total of 8 weeks.
  Arms: Sham excimer laser

SUMMARY:
Psoriasis is a common skin disease, which affects 2-3% of the population. Up to two third of patients with psoriasis develop nail changes. These visible changes can be painful and disabling and are associated with social stigma. Most topical treatments are only partially effective. Systemic treatments can have serious side effects. Excimer laser is a form of targeted ultraviolet light therapy that has been successfully used to treat isolated psoriatic plaques on difficult to treat areas such as scalp or palms. The purpose of this study is to investigate efficacy of excimer laser for treatment of fingernail psoriasis. Sixteen patients with stable fairly symmetric fingernail psoriasis will be enrolled. After obtaining informed consent, an investigator will evaluate the severity of nail psoriasis in each hand using an objective score, called Modified Nail Psoriasis Severity Index (mNAPSI). In a random fashion, one hand will be treated with excimer laser and the other hand will receive sham treatment. During the treatments, patients will wear protective eyewear that does not permit them to see which hand receives active treatment and which hand receives sham treatment. Patients will be treated twice a week for 8 weeks. At weeks 8, 12, and16 the investigator who is blinded to the treatment assignments will re-evaluate the fingernails using mNAPSI score. Mean change from baseline mNAPSI score at weeks 8, 12, and 16 in hands treated with excimer compared to hands treated with sham will be measured. We will also measure patient's assessment of severity of nail disease and the pain or any adverse events associated with laser treatments. Given the slow growth rate of fingernails, the final evaluations will be performed at week 16. In summary, this is the first controlled study to evaluate efficacy of excimer laser in fingernail psoriasis. If found to be effective, excimer laser could be used as a safe, locally administered treatment for recalcitrant nail psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent.
* Must be at least 18 years old.
* Must have been diagnosed with stable fingernail psoriasis.
* Must have fairly symmetric fingernail psoriasis in right and left hand with similar modified NAPSI scores in right and left hand target nails. Target nail is defined as the fingernail with highest modified NAPSI score.
* Must have active fingernail psoriasis, defined as a target fingernail matrix NAPSI score of at least 2 and modified NAPSI score from a combination of crumbling, onycholysis and pitting at least 2. •
* No changes in the systemic therapy or nail directed topical therapy during the 16 week study period.

Exclusion criteria:

* Subjects unable to tolerate frequency of visits.
* History of intolerance to or worsening of psoriasis with ultraviolet light.
* Current use of known photosensitizing medications.
* History of Fitzpatrick Type I skin, photosensitivity, or keloid formation.
* Any new systemic psoriasis therapy including biologics, conventional systemic immunomodulators, phototherapy, or nail directed topical therapy for the last 3 months prior to enrollment.
* Any other condition that in the eyes of the investigator will disqualify patient from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Department of Dermatology, Salt Lake City, Utah, United States

REFERENCES:
- [Background] Augustin M, Herberger K, Hintzen S, Heigel H, Franzke N, Schafer I. Prevalence of skin lesions and need for treatment in a cohort of 90 880 workers. Br J Dermatol. 2011 Oct;165(4):865-73. doi: 10.1111/j.1365-2133.2011.10436.x. PMID 21623753
- [Background] Schafer I, Rustenbach SJ, Radtke M, Augustin J, Glaeske G, Augustin M. [Epidemiology of psoriasis in Germany--analysis of secondary health insurance data]. Gesundheitswesen. 2011 May;73(5):308-13. doi: 10.1055/s-0030-1252022. Epub 2010 Jun 11. German. PMID 20544588
- [Background] de Jong EM, Seegers BA, Gulinck MK, Boezeman JB, van de Kerkhof PC. Psoriasis of the nails associated with disability in a large number of patients: results of a recent interview with 1,728 patients. Dermatology. 1996;193(4):300-3. doi: 10.1159/000246274. PMID 8993953
- [Background] Klaassen KM, van de Kerkhof PC, Pasch MC. Nail psoriasis: a questionnaire-based survey. Br J Dermatol. 2013 Aug;169(2):314-9. doi: 10.1111/bjd.12354. PMID 23550612
- [Background] van der Velden HM, Klaassen KM, van de Kerkhof PC, Pasch MC. Fingernail psoriasis reconsidered: a case-control study. J Am Acad Dermatol. 2013 Aug;69(2):245-52. doi: 10.1016/j.jaad.2013.02.009. Epub 2013 Mar 28. PMID 23541759
- [Background] de Vries AC, Bogaards NA, Hooft L, Velema M, Pasch M, Lebwohl M, Spuls PI. Interventions for nail psoriasis. Cochrane Database Syst Rev. 2013 Jan 31;2013(1):CD007633. doi: 10.1002/14651858.CD007633.pub2. PMID 23440816
- [Background] Marx JL, Scher RK. Response of psoriatic nails to oral photochemotherapy. Arch Dermatol. 1980 Sep;116(9):1023-24. PMID 7416754
- [Background] [Narrow spectrum (311 nm) phototherapy in treatment of psoriatic nail]. Georgian Med News. 2009 Feb;(167):56-9. Russian. PMID 19276472
- [Background] Aubin F, Vigan M, Puzenat E, Blanc D, Drobacheff C, Deprez P, Humbert P, Laurent R. Evaluation of a novel 308-nm monochromatic excimer light delivery system in dermatology: a pilot study in different chronic localized dermatoses. Br J Dermatol. 2005 Jan;152(1):99-103. doi: 10.1111/j.1365-2133.2005.06320.x. PMID 15656808
- [Background] Mudigonda T, Dabade TS, Feldman SR. A review of protocols for 308 nm excimer laser phototherapy in psoriasis. J Drugs Dermatol. 2012 Jan;11(1):92-7. PMID 22206083
- [Background] Mudigonda T, Dabade TS, West CE, Feldman SR. Therapeutic modalities for localized psoriasis: 308-nm UVB excimer laser versus nontargeted phototherapy. Cutis. 2012 Sep;90(3):149-54. PMID 23094316
- [Background] Al-Mutairi N, Al-Haddad A. Targeted phototherapy using 308 nm Xecl monochromatic excimer laser for psoriasis at difficult to treat sites. Lasers Med Sci. 2013 Jul;28(4):1119-24. doi: 10.1007/s10103-012-1210-4. Epub 2012 Sep 28. PMID 23053247
- [Background] Asawanonda P, Anderson RR, Chang Y, Taylor CR. 308-nm excimer laser for the treatment of psoriasis: a dose-response study. Arch Dermatol. 2000 May;136(5):619-24. doi: 10.1001/archderm.136.5.619. PMID 10815855
- [Background] Rich P, Scher RK. Nail Psoriasis Severity Index: a useful tool for evaluation of nail psoriasis. J Am Acad Dermatol. 2003 Aug;49(2):206-12. doi: 10.1067/s0190-9622(03)00910-1. PMID 12894066
- [Background] Aktan S, Ilknur T, Akin C, Ozkan S. Interobserver reliability of the Nail Psoriasis Severity Index. Clin Exp Dermatol. 2007 Mar;32(2):141-4. doi: 10.1111/j.1365-2230.2006.02305.x. Epub 2006 Nov 27. PMID 17137477
- [Background] Cassell SE, Bieber JD, Rich P, Tutuncu ZN, Lee SJ, Kalunian KC, Wu CW, Kavanaugh A. The modified Nail Psoriasis Severity Index: validation of an instrument to assess psoriatic nail involvement in patients with psoriatic arthritis. J Rheumatol. 2007 Jan;34(1):123-9. PMID 17216680
- [Background] Yaemsiri S, Hou N, Slining MM, He K. Growth rate of human fingernails and toenails in healthy American young adults. J Eur Acad Dermatol Venereol. 2010 Apr;24(4):420-3. doi: 10.1111/j.1468-3083.2009.03426.x. Epub 2009 Sep 8. PMID 19744178
- [Background] Ortonne JP, Paul C, Berardesca E, Marino V, Gallo G, Brault Y, Germain JM. A 24-week randomized clinical trial investigating the efficacy and safety of two doses of etanercept in nail psoriasis. Br J Dermatol. 2013 May;168(5):1080-7. doi: 10.1111/bjd.12060. PMID 23013207
- [Background] de Jong EM, Menke HE, van Praag MC, van De Kerkhof PC. Dystrophic psoriatic fingernails treated with 1% 5-fluorouracil in a nail penetration-enhancing vehicle: a double-blind study. Dermatology. 1999;199(4):313-8. doi: 10.1159/000018281. PMID 10640840

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: all participants received 308 nm excimer laser treatment on one hand, and sham laser treatment on the other hand
  308 nm excimer laser: Biweekly treatments with 308 nm excimer laser for a total of 8 weeks
Period: Overall Study
Arm/Group | All Study Participants
Started | 8
Completed | 7
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: all study participants received 308 nm excimer laser treatment to one hand and sham laser to the other hand.
  308 nm excimer laser: Biweekly treatments with 308 nm excimer laser for a total of 8 weeks
Arm/Group | All Study Participants
Number analyzed (Participants) | 8
Age, Continuous [Mean (Full Range); unit: years] | 45 [19 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Modified NAPSI Score (Nail Psoriasis Severity Index)
Description: This is an instrument that scores nail psoriasis severity. Severity for each nail is measured on a scale of 0-13, where crumbling, pitting, onycholysis and oil spots together are each graded 0-3, and other features (leukonychia, splinter hemorrhages, hyperkeratosis, and red spots in lunula) are scored 0 (absent) or 1 (present). Higher score indicates more severe nail psoriasis with 13 being the most severe and 0 being no nail disease present.
Time Frame: at 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active: 308 nm excimer laser treatment
  308 nm excimer laser: Biweekly treatments with 308 nm excimer laser for a total of 8 weeks
  308 nm excimer laser: Laser to the non-control side
- Sham: Sham laser treatment.
  Sham laser: Biweekly treatments with Sham laser for a total of 8 weeks.
  Sham laser: Sham laser treatment to the control side (308 nm excimer laser with cover in place preventing patient from exposure to laser energy).
Arm/Group | Active | Sham
Number analyzed (Participants) | 7 | 7
units on a scale | 6.3 (1.8) | 6.0 (1.3)

2. Secondary Outcome: Patient Assessment of Nail Psoriasis Activity
Description: this is a subjective patient reported scale, 0-100, where 100 is the most severe global assessment of the patient's nail psoriasis, and 0 is clear (no nail disease present).
Time Frame: at 16 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Active: 308 nm excimer laser treatment
  308 nm excimer laser: Biweekly treatments with 308 nm excimer laser for a total of 8 weeks
- Sham: Sham 308 nm excimer laser treatment
  Sham laser: Sham laser treatment to the control side.
Arm/Group | Active | Sham
Number analyzed (Participants) | 7 | 7
units on a scale | 58.6 (33.0) | 55.4 (24.3)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 16 weeks (entire time of participation for each subject from screening to termination.
Groups:
- Sham: Sham laser treatment (laser covered with cap so that the patient is not exposed to laser energy)
  Sham laser: Biweekly treatments with Sham laser for a total of 8 weeks
Arm/Group | Active | Sham
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes